CLINICAL TRIAL: NCT05105841
Title: A Phase 2 Study of the Safety and Efficacy of Venetoclax in Combination With Obinutuzumab or Ibrutinib in Japanese Subjects With Previously Untreated Chronic Lymphocytic Leukemia (CLL)/Small Lymphocytic Lymphoma (SLL)
Brief Title: Study to Assess Change in Disease Activity and Adverse Events of Oral Venetoclax in Combination With Intravenous (IV) Obinutuzumab or Oral Ibrutinib in Adult Participants With Untreated Chronic Lymphocytic Leukemia (CLL)/Small Lymphocytic Lymphoma (SLL)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: M20-353
Expanded Access: NCT03123029 (Available)
Record Dates: First submitted 2021-10-25; First posted 2021-11-03 (Actual); Last update posted 2025-10-15 (Actual); Status verified 2025-08

CONDITIONS: Chronic Lymphocytic Leukemia (CLL); Small Lymphocytic Lymphoma (SLL)
Keywords: Chronic Lymphocytic Leukemia (CLL); Small Lymphocytic Lymphoma (SLL); Ibrutinib; Imbruvica; Venetoclax; Venclexta; Venclyxto; Obinutuzumab; GA101; Gazyva; RO5072759
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell | interventions — venetoclax; ibrutinib; obinutuzumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Venetoclax + Obinutuzumab (V+G) (Experimental): Participants will receive venetoclax + obinutuzumab for twelve 28-day cycles.
  Interventions: Drug: Venetoclax; Drug: Obinutuzumab
- Venetoclax + Ibrutinib (V+I) (Experimental): Participants will receive venetoclax + ibrutinib for fifteen 28-day cycles.
  Interventions: Drug: Venetoclax; Drug: Ibrutinib

INTERVENTIONS:
Drug: Venetoclax — Oral Tablet
  Other Names: Venclexta; ABT-199; GDC-0199
Drug: Ibrutinib — Oral Capsule
  Other Names: Imbruvica
  Arms: Venetoclax + Ibrutinib (V+I)
Drug: Obinutuzumab — Intravenous (IV) Infusion
  Other Names: GA101; Gazyva; RO5072759
  Arms: Venetoclax + Obinutuzumab (V+G)

SUMMARY:
Chronic lymphocytic leukemia (CLL) is the most common leukemia in Western countries, representing approximately 30% of all adult leukemias. There is a large difference in proportion of malignant lymphoma between the United States (US) and Japan was seen in CLL/small lymphocytic lymphoma (SLL) (Japan, 3.2%; US, 24.1%). The purpose of this study is to assess how well venetoclax works in combination with obinutuzumab (V+G, Cohort 1) or with ibrutinib (V+I, Cohort 2) in Japanese participants with previously untreated CLL/Small Lymphocytic Lymphoma (SLL). Adverse events and change in disease activity will be assessed.

Venetoclax is an approved drug for the treatment of CLL and SLL. Study doctors put the participants in 1 of 2 groups, called treatment arms, based on variable alternating assignment. Approximately 20 adult participants with previously untreated CLL/SLL will be enrolled in the study in approximately 20 sites in Japan.

Participants in group 1 will receive oral venetoclax + intravenous (IV) obinutuzumab (V+G) in 28-day cycles for a total of 12 cycles, and participants in group 2 will receive oral venetoclax + oral ibrutinib (V+I) in 28-day cycles for a total of 15 cycles.

There may be higher treatment burden for participants in this trial compared to their standard of care. Participants will attend regular visits during the study at a hospital or clinic. The effect of the treatment will be checked by medical assessments, blood tests, and checking for side effects.

ELIGIBILITY:
Inclusion Criteria:

* Adult male or female, at least ≥ 65 years old; or 20 to 64 years old and have at least 1 of the following:

  * Cumulative Illness Rating Scale (CIRS) score > 6.
  * Creatinine clearance (CrCl) estimated < 70 mL/min using Cockcroft-Gault equation.
* Must have measurable nodal disease (by computed tomography [CT]), defined as at least one lymph node > 1.5 cm in longest diameter.
* Diagnosed Chronic Lymphocytic Leukemia (CLL)/Small Lymphocytic Lymphoma (SLL) that requires treatment according to the Modified 2008 International Workshop on Chronic Lymphocytic Leukemia (iwCLL) criteria.

Exclusion Criteria:

* Transformation of Chronic Lymphocytic Leukemia (CLL) to aggressive non-Hodgkin lymphoma (NHL; Richter's transformation or pro-lymphocytic leukemia).
* Previous treatment history for CLL/SLL.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2021-11-08 (Actual); Primary Completion 2025-10-09 (Actual); Study Completion 2025-10-09 (Actual)

PRIMARY OUTCOMES:
Complete Remission (CR) with an Incomplete Marrow Recovery (CRi) Rate, as Assessed by an Independent Review Committee (IRC) per Modified 2008 International Workshop on Chronic Lymphocytic Leukemia (iwCLL) for Venetoclax + Obinutuzumab (V+G) | Up to Week 32
  CR rate is defined as the percentage of participants achieving a best response of CR or CRi.
CR/CRi Rate, as Assessed by an IRC per iwCLL for Venetoclax + Ibrutinib (V+I) | Up to Week 56
  CR rate is defined as the percentage of participants achieving a best response of CR or CRi.

SECONDARY OUTCOMES:
CR/CRi Rate, as Assessed by an Investigator per iwCLL for (V+G) | Up to Week 32
  CR rate is defined as the percentage of participants achieving a best response of CR or CRi.
CR/CRi Rate, as Assessed by an Investigator per iwCLL for (V+I) | Up to Week 56
  CR rate is defined as the percentage of participants achieving a best response of CR or CRi.
Overall response rate (ORR) as Assessed by IRC for (V+G) | Up to Week 32
  ORR is defined as the proportion of participants with a best overall response of CR, CRi, partial remission (PR) or nodular partial remission (nPR) per 2008 iwCLL criteria as assessed by an IRC.
ORR as Assessed by IRC (V+I) | Up to Week 56
  ORR is defined as the proportion of participants with a best overall response of CR, CRi, partial remission (PR) or nodular partial remission (nPR) per 2008 iwCLL criteria as assessed by an IRC.
ORR as Assessed by Investigator for (V+G) | Up to Week 32
  ORR is defined as the proportion of participants with a best overall response of CR, CRi, partial remission (PR) or nodular partial remission (nPR) per 2008 iwCLL criteria as assessed by an investigator.
ORR Assessed by Investigator + Ibrutinib (V+I) | Up to Week 56
  ORR is defined as the proportion of participants with a best overall response of CR, CRi, partial remission (PR) or nodular partial remission (nPR) per 2008 iwCLL criteria as assessed by an investigator.
Progression-Free Survival (PFS) as Assessed by IRC for (V+G) | Up to Week 32
  PFS is defined as the time from the date of first dose of any study drug until the date of disease progression or death due to any cause, whichever occurs first, as determined by an IRC according to iwCLL criteria.
PFS as Assessed by IRC for (V+I) | Up to Week 56
  PFS is defined as the time from the date of first dose of any study drug until the date of disease progression or death due to any cause, whichever occurs first, as determined by an IRC according to iwCLL criteria.
PFS as Assessed by Investigator for (V+G) | Up to Week 32
  PFS is defined as the time from the date of first dose of any study drug until the date of disease progression or death due to any cause, whichever occurs first, as determined by an investigator according to iwCLL criteria.
PFS as Assessed by Investigator for (V+I) | Up to Week 56
  PFS is defined as the time from the date of first dose of any study drug until the date of disease progression or death due to any cause, whichever occurs first, as determined by an investigator according to iwCLL criteria.
Duration of response (DOR) as Assessed by IRC for (V+G) | Up to Week 32
  DOR is defined as the time from the first occurrence of overall response (CR, CRi, PR or nPR) until disease progression or death due to any cause, whichever occurs first, as determined by an IRC according to iwCLL criteria.
DOR as Assessed by IRC for (V+I) | Up to Week 56
  DOR is defined as the time from the first occurrence of overall response (CR, CRi, PR or nPR) until disease progression or death due to any cause, whichever occurs first, as determined by an IRC according to iwCLL criteria.
DOR as Assessed by Investigator for (V+G) | Up to Week 32
  DOR is defined as the time from the first occurrence of overall response (CR, CRi, PR or nPR) until disease progression or death due to any cause, whichever occurs first, as determined by an investigator according to iwCLL criteria.
DOR as Assessed by Investigator for (V+I) | Up to Week 56
  DOR is defined as the time from the first occurrence of overall response (CR, CRi, PR or nPR) until disease progression or death due to any cause, whichever occurs first, as determined by an investigator according to iwCLL criteria.
Overall Survival (OS) for (V+G) | Up to Week 32
  OS is defined as the time from the date of the first dose of any study drug until death due to any cause.
OS for (V+I) | Up to Week 56
  OS is defined as the time from the date of the first dose of any study drug until death due to any cause.
Time to progression (TTP) as Assessed by IRC for (V+G) | Up to Week 32
  TTP is defined as the time from the date of first dose of any study drug until the date of disease progression, as determined by an IRC according to iwCLL criteria.
TTP as Assessed by IRC for (V+I) | Up to Week 56
  TTP is defined as the time from the date of first dose of any study drug until the date of disease progression, as determined by an IRC according to iwCLL criteria.
TTP as Assessed by Investigator for (V+G) | Up to Week 32
  TTP is defined as the time from the date of first dose of any study drug until the date of disease progression, as determined by an investigator according to iwCLL criteria.
TTP as Assessed by Investigator for (V+I) | Up to Week 56
  TTP is defined as the time from the date of first dose of any study drug until the date of disease progression, as determined by an investigator according to iwCLL criteria.

CONTACTS AND LOCATIONS:
Overall Officials: ABBVIE INC., Study Director — AbbVie
Locations (20):
- Japan (20):
  - Duplicate_NHO Nagoya Medical Center /ID# 233523, Nagoya, Aichi-ken
  - Aichi Cancer Center Hospital /ID# 238797, Nagoya, Aichi-ken
  - Duplicate_Japanese Red Cross Aichi Medical Center Nagoya Daini Hospital /ID# 233524, Nagoya, Aichi-ken
  - Duplicate_Chiba Cancer Center /ID# 238839, Chiba, Chiba
  - National Hospital Organization Shikoku Cancer Center /ID# 234059, Matsuyama, Ehime
  - Kyushu University Hospital /ID# 238437, Fukuoka, Fukuoka
  - Duplicate_Hokkaido University Hospital /ID# 238377, Sapporo, Hokkaido
  - Hyogo Prefectural Amagasaki General Medical Center /ID# 234082, Amagasaki-shi, Hyōgo
  - Tokai University Hospital /ID# 238970, Isehara, Kanagawa
  - University Hospital Kyoto Prefectural University of Medicine /ID# 239883, Kyoto, Kyoto
  - Tohoku University Hospital /ID# 238433, Sendai, Miyagi
  - Niigata University Medical & Dental Hospital /ID# 238324, Niigata, Niigata
  - Duplicate_Okayama University Hospital /ID# 238467, Okayama, Okayama-ken
  - Kindai University Hospital /ID# 234001, Osakasayama-shi, Osaka
  - Duplicate_Osaka University Hospital /ID# 234037, Suita-shi, Osaka
  - Duplicate_Shimane University Hospital /ID# 234076, Izumo-shi, Shimane
  - Duplicate_Jichi Medical University Hospital /ID# 238434, Shimotsuke-shi, Tochigi
  - National Cancer Center Hospital /ID# 232449, Chuo-ku, Tokyo
  - The Cancer Institute Hospital Of JFCR /ID# 232450, Koto-ku, Tokyo
  - Yamagata University Hospital /ID# 234032, Yamagata, Yamagata

IPD SHARING:
Plan to Share IPD: Yes
AbbVie is committed to responsible clinical trial data sharing. This includes access to anonymized, individual and trial-level data (analysis data sets), as well as other information.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: For details on when studies are available for sharing visit https://vivli.org/ourmember/abbvie/
Access Criteria: To learn more about the process, or to submit a request, visit the following link https://www.abbvieclinicaltrials.com/hcp/data-sharing/
URL: https://vivli.org/ourmember/abbvie/

REFERENCES:
- See also: Related info — https://www.rxabbvie.com/